CLINICAL TRIAL: NCT03945838
Title: Assessment of Muscle Strength and Volume Changes in Patients With Breast Cancer- Related Lymphedema
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Göksel Tanıgör M.D., Researcher in Ege University School of Medicine, Ege University
Other Study IDs: LymphHG
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Lymphedema Arm; Lymphedema; Surgical
Keywords: Lymphedema; Hand grip strength; Breast cancer related lymphedema; Complete decongestion therapy
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer related lymphedema: All patients were included in the complete decongestive therapy programme. This therapy includes patient education, skin care, exercises, manual lymphatic drainage (self), and compression bandage therapy.
  Interventions: Other: Complete Decongestion Therapy

INTERVENTIONS:
Other: Complete Decongestion Therapy — It is given in two phases. First phase includes intensive therapy which aims to reduce the volume of the extremity. Second phase aims to preserve these reductions of volume.
  All patients were prescribed lymphedema specific exercises and were advised to walk (for 30 minutes everyday) daywhile taking complete decongestive therapy. They were specifically informed that exercise does not aggravate the severity of their lymphedema.
  Short stretch bandages were applied to the patients with self manual lymphatic drainage. Intensive phase was given 5 days a week, and short stretch bandages applied for 23 hours a day with 1 hour interval. To increase the local pressure on the areas required, foams were added. Patients were screened with arm circumferential measurements once a week. After gaining a plateau in the volumes, patients were prescribed compression garments.

SUMMARY:
This study aims to find whether complete decongestive therapy used in breast cancer-related lymphedema has an effect on muscle strength in the affected arm, while assessing the efficacy of the therapy itself. 74 patients with breast cancer related lymphedema were included in this study. Patients were taken their demographic and clinical history and were evaluated with measurements of extremity volumes and hand grip strengths using a hand dynamometer before and after the complete decongestive therapy. Data were then assessed using relevant statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Having had mastectomy or breast conserving surgery
* Having a certain diagnosis of lymphedema with a difference in arm circumferences more than 1 cm

Exclusion Criteria:

* The subjects with active infection or cancer with metastases, the ones who didn't accept the complete decongestive therapy, patients with vascular disease, rheumatic disease, upper limb deformity, any upper limb surgery history, bilateral lymphedema or a history of transplantation were excluded

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18-70 years old with a history of mastectomy or breast conserving surgery and lymphedema
  * Having a certain diagnosis of lymphedema
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 3 weeks
  Hand grip strength: Hand grip strength was measured using JAMAR® hand dynamometer. It has been used to assess hand grip strength in many studies over half a century. Patients were asked to sit down with shoulder adducted, elbow flexed (90°) and forearm in the neutral position. Mean of the 3 measurements taken with 1 minute apart from each other was recorded. Patients' measurements were taken for both affected and unaffected arm, and recorded as kgf.
Extremity volume | 3 weeks
  Volume measurements were taken using ulnar styloid process as a index point, and circumferential measurements were taken with 5 cm spaces from distal to the proximal. Using a computer programme (Limb Volumes Professional version 5.0), the total volume of the arm was calculated and recorded before and after the treatment for both arms.
  All patients' measurements were taken by the same researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university school of medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No